CLINICAL TRIAL: NCT05213637
Title: A Multicenter, Randomized, Open-label Phase II Study of Expanded Activated Lymphocytes (EAL) as Adjuvant Therapy in Preventing Recurrence in Patients With Primary Hepatocellular Carcinoma (HCC) at High Recurrence Risk After Radical Resection
Brief Title: Expanded Activated Lymphocytes (EAL) as Adjuvant Therapy in Patients With HCC at High Risk of Recurrence After Radical Resection
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Immunotech Applied Science Ltd. (Industry)
Responsible Party: Principal Investigator, Prof. Shichun Lu, Director, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EAL-HCC-001
Record Dates: First submitted 2022-01-27; First posted 2022-01-28 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: HCC; cell therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EAL Treatment Group (Experimental): The patients with primary HCC will receive 12~20 doses of EAL infusion (1×10^9~2×10^10 cells per dose) in combination of a single transarterial chemoembolization (TACE) after radical resection.
  Interventions: Biological: Expanded Activated Lymphocytes (EAL); Procedure: transarterial chemoembolization (TACE)
- Control Group (Active Comparator): The patients with primary HCC will receive a single TACE after radical resection.
  Interventions: Procedure: transarterial chemoembolization (TACE)

INTERVENTIONS:
Biological: Expanded Activated Lymphocytes (EAL) — 12~20 doses of EAL (1×10^9~2×10^10 cells per dose) will be infused into patients.
  Arms: EAL Treatment Group
Procedure: transarterial chemoembolization (TACE) — After angiography, fluorouracil will be injected into the proper hepatic artery or the segment of liver where the original lesion is located, and then microcatheter will be introduced into the segment of liver artery where the incision margin is located, and iodized oil injection and epirubicin will be mixed and embolized.

SUMMARY:
This is a multi-center, randomized, open-label pivotal phase II study to evaluate the efficacy and safety of EAL as adjuvant therapy in preventing recurrence in patients with primary HCC at high recurrence risk after radical resection.

DETAILED DESCRIPTION:
HCC, accounting for 80% of all liver cancers, is the third most common cause of cancer-related death worldwide. Radical resection is considered as a curative strategy for patients with primary HCC. However, over 50% of patients experience recurrence after resection, resulting in a very low 5-year survival rate. EAL are ex vivo expanded and activated lymphocytes comprising mainly CD8+ T cells derived from patients' peripheral blood. This is a multi-center, randomized, open-label pivotal phase II study to evaluate the efficacy and safety of EAL in preventing recurrence in patients with primary HCC at high recurrence risk after radical resection. Patients will be randomized in a 1:1 ratio to receive either 20 doses of EAL (1×10^9~2×10^10 per dose) infusion in combination of a single TACE or a single TACE only. Primary endpoint is the independent review committee-determined recurrence-free survival (from randomization to first recurrence or death from any cause). Secondary endpoints include overall survival, cancer-specific survival, adverse events and others.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Stage Ia~IIIa primary HCC with high recurrence risk (defined as single tumor ≥5cm in diameter, or single tumor <5cm in diameter with MVI, PVTT, hepatic vein invasion, satellite lesions or AFP ≥400ng/mL, or multiple tumors).
2. Patients who have undergone a radical resection.
3. ECOG PS Score 0~2.
4. Child-Pugh Score ≤ 7.
5. Patients with adequate hematologic and end-organ function.
6. HBV-HCC and HCV-HCC patients with active viral infection may receive antiviral treatment simultaneously.
7. Patients who have a life expectancy of at least 6 months.

Exclusion Criteria:

1. Patients with a history of immune deficiency or autoimmune diseases (such as rheumatoid joint disease, systemic lupus erythematosus, vasculitis, multiple sclerosis, insulin-dependent diabetes mellitus, etc.).
2. Patients with a history of other malignant tumors in the past 5 years.
3. Patients who received chemotherapy, radiotherapy, molecular targeted therapy, biological immunotherapy, and hormone therapy within 1 month prior to screening.
4. Patients who have received microwave ablation, cryotherapy, high-power ultrasound focused ablation and other local ablation methods for liver tumors.
5. Patients with postoperative organ dysfunction or heart and lung diseases.
6. Patients allergic to albumin or with serious allergy history or mental disease.
7. Pregnant or lactating women.
8. Anticipated other clinical trials within 4 weeks before this trial.
9. Patients with HIV or Treponema pallidum infection, septicemia and other uncontrolled infection.
10. Patients after organ or bone marrow transplant.
11. Patients with drug or alcohol abuse/addiction.
12. Any condition that would, in the investigator's judgment, make it unsuitable for the donors to be enrolled.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2018-04-25 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival (RFS) | 6 years
  The time from randomization to first documented of disease recurrence determined by IRC or death from any cause (whichever occurs first).

SECONDARY OUTCOMES:
Overall survival (OS) | 6 years
  The time from randomization to death from any cause.
Cancer-specific survival (CSS) | 6 years
  The time from randomization to death from HCC.
Adverse events (AE) | 6 years
  Percentage of participants with adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Shichun Lu, MD, PhD, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China